CLINICAL TRIAL: NCT01019941
Title: Open Label, Randomized, Single-dose, Crossover Study to Evaluate the Pharmacokinetics of Docetaxel Between Two Docetaxel Products, CKD-810 and Taxotere Inj., in Patients With Advanced Solid Cancer
Brief Title: Pharmacokinetic Study of CKD-810 and Taxotere to Treat Patient With Advanced Solid Cancer
Acronym: 126ASC08Q
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Jin Kim, Chong Kun Dang
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CKD-810_PK_phase I
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Advanced Solid Cancers
Keywords: Docetaxel; CKD-810; Taxotere inj.; Advanced Solid cancer; Pharmacokinetic evaluation
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1st cycle:CKD-810 -> 2nd cycle:Taxotere inj. (Other)
  Interventions: Drug: CKD-810, Taxotere inj.
- 1st cycle:Taxotere inj.-> 2nd cycle:CKD-810 (Other)
  Interventions: Drug: CKD-810, Taxotere inj.

INTERVENTIONS:
Drug: CKD-810, Taxotere inj. — Patients will receive docetaxel 75mg/㎡ on Day 1 of each cycle(1 cycle = 3 weeks) as a 1-hour IV infusion. At the 1st cycle, CKD-810 75mg/㎡ administered. If the hematologic or non-hematologic toxicity was not appeared when the 1st cycle intervention was finished, keep going the 2nd cycle intervention.
  Other Names: Docetaxel anhydrous, Docetaxel
  Arms: 1st cycle:CKD-810 -> 2nd cycle:Taxotere inj.
Drug: CKD-810, Taxotere inj. — Patients will receive docetaxel 75mg/㎡ on Day 1 of each cycle(1 cycle = 3 weeks) as a 1-hour IV infusion. At the 1st cycle, Taxotere inj. 75mg/㎡ administered. If the hematologic or non-hematologic toxicity was not appeared when the 1st cycle intervention was finished, keep going the 2nd cycle intervention.
  Other Names: Docetaxel anhydrous, Docetaxel
  Arms: 1st cycle:Taxotere inj.-> 2nd cycle:CKD-810

SUMMARY:
The purpose of this study is to evaluate safety and the pharmacokinetic characteristics of docetaxel between two docetaxel products in patients with advanced solid cancer.

DETAILED DESCRIPTION:
This is a Phase III study designed to evaluate the pharmacokinetic characteristics of docetaxel between two docetaxel products in patients with advanced solid cancer. This study will also assess the safety of the docetaxel in advanced solid cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is greater than 18 years of age
* Advanced solid tumor

  * locally advanced or metastatic breast cancer which docetaxel alone therapy was adequate
  * locally advanced or metastatic non-small cell lung cancer which docetaxel alone therapy was adequate
  * locally advanced or metastatic other malignant tumor which docetaxel alone therapy was adequate
* Patient has a life expectancy of at least 3 months
* Patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Absolute neutrophil count ≥ 1,500/㎣
* Platelet count ≥ 100,000/㎣
* Hemoglobin ≥ 9.0g/dL
* Total Bilirubin ≤ 1.5 X ULN
* Alkaline Phosphatase ≤ 2.5 X ULN
* AST/ALT ≤ 2.0 X ULN
* Serum creatinine ≤ 1.5 X ULN or Creatinine clearance ≥ 60mL/min(Cockcroft equation)
* Patients should voluntarily sign a written informed consent before study entry

Exclusion Criteria:

* If present, any active bacterial infection that have to parenteral antibiotic therapy. Patients may be included if their infection has resolved to totally or controlled state
* Brain metastasis with neurologic symptom
* History of unstable cardiac arrhythmia, congestive heart failure or myocardial infarction within 6 months
* Known to test positive for HIV or hepatitis B or C
* Use of inducers or inhibitors of CYP3A4 within 2 weeks prior to the first dose of study medication. (Patients may be included if the patients who need to intake the medication such as cimetidine was keep the same dose continuously at 1 cycle and 2 cycle)
* Peripheral neuropathy ≥ Grade 2
* known resistant or uncontrolled severe hypersensitivity to docetaxel
* History of hypersensitivity reaction to Polysorbate 80
* The female patients of pregnancy, breast feeding or childbearing potential. And the patients has not laboratory result or the result was a positive serum pregnancy test, also Patients (M/F) with reproductive potential not implementing adequate contraceptive measurements. (In case of menopausal women, keeping menopause at least 12 months. All sexually active male patients must agree to use adequate methods of birth control throughout the study)
* Administration of any other tumor therapy, including chemotherapy, radiotherapy, and immunotherapy within 4 weeks before the beginning of study treatment. Patients may be included if the radiotherapy was conducted to relieve symptoms and that symptoms recovered to grade 1
* treated with any investigational drugs within 4 weeks before the beginning of study treatment
* Must be treated concurrent administration of other anti-cancer medicine
* Not able to participate to the study, at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of CKD-810 and Taxotere inj. | 2 Cycles

SECONDARY OUTCOMES:
Safety of CKD-810 and Taxotere inj. | 2 Cycles

CONTACTS AND LOCATIONS:
Overall Officials: JH Kang, Principal Investigator — The Catholic University of Korea
Locations (7):
- South Korea (7):
  - Gachon University Gil Hospital, Inchon
  - The Catholic university of KOREA, Seoul ST. Mary's Hospital, Seoul
  - The Korea University Anam Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Dongsan Medical Center, Keimyung University, Taegu
  - Yeoungnam University Hospital, Taegu
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Cho EK, Park JY, Lee KH, Song HS, Min YJ, Kim YH, Kang JH. Open-label, randomized, single-dose, crossover study to evaluate the pharmacokinetics and safety differences between two docetaxel products, CKD-810 and Taxotere injection, in patients with advanced solid cancer. Cancer Chemother Pharmacol. 2014 Jan;73(1):9-16. doi: 10.1007/s00280-013-2264-0. Epub 2013 Dec 12. PMID 24337589